CLINICAL TRIAL: NCT06511141
Title: Sacral Neuromodulation for Male Overactive Bladder
Brief Title: Sacral Neuromodulation for Male Overactive Bladder (MOAB)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Axonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105-0141
Record Dates: First submitted 2024-07-16; First posted 2024-07-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Overactive Bladder; Urinary Urgency Incontinence; Benign Prostatic Hyperplasia; Prostate Cancer; Prostatectomy; Urinary Frequency
MeSH Terms: conditions — Urinary Bladder, Overactive; Prostatic Hyperplasia; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Post-prostatectomy (Other): History of radical prostatectomy for cancer treatment at least 6 months prior to enrollment
  Interventions: Device: Axonics SNM System
- Radiation (Other): History of radiation for cancer treatment at least 6 months prior to enrollment
  Interventions: Device: Axonics SNM System
- Benign Prostatic Hyperplasia (BPH) (Other): History of cytoreductive BPH surgery at least 6 months prior to enrollment
  Interventions: Device: Axonics SNM System

INTERVENTIONS:
Device: Axonics SNM System — To assess clinical outcomes of the Axonics SNM System in the male OAB population.

SUMMARY:
To assess the post-market clinical outcomes of the Axonics SNM System for treatment of overactive bladder in male patients.

DETAILED DESCRIPTION:
To assess the post-market clinical outcomes of the Axonics SNM System for treatment of overactive bladder in male patients who have a prior history of radical prostatectomy or radiation for prostate cancer or who have a history of cytoreductive surgical intervention for benign prostatic hyperplasia (BPH).

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants aged ≥ 18 years at the time of enrollment
2. Able to complete bladder diaries and patient questionnaires
3. Primary diagnosis of OAB (urinary urgency incontinence (UUI) or urinary frequency (UF)).
4. Willing and capable to provide written informed consent and agrees to comply with specified evaluations at clinical investigational sites and attend all follow-up assessments for up to 1 year

Key Exclusion Criteria:

1. Any patient that is not a suitable candidate per investigator discretion
2. Recent prostate therapy or procedure within the last 6 months at the time of enrollment
3. Any neurological condition that could interfere with normal bladder function, including stroke, epilepsy, multiple sclerosis, Parkinson's disease, clinically significant peripheral neuropathy, or spinal cord injury (e.g., paraplegia)
4. Previously implanted with a sacral neuromodulation device, including inactive SNM devices
5. Any prior treatment with an Implantable Tibial Nerve Stimulation (ITNS)
6. Positive response to Percutaneous Tibial Nerve Stimulation (PTNS) within the last 3 months at the time of enrollment
7. Underwent an external trial with any sacral neuromodulation device and was deemed a non-responder by a physician
8. Any significant medical condition that is likely to interfere with study procedures, device operation, or likely to confound evaluation of study objectives at the discretion of the participating physician.
9. Uncontrolled diabetes
10. Known allergic reactions to components of the Axonics SNM System, including titanium, zirconia, polyurethane, epoxy, or silicone

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male patients will be enrolled in this study.
Enrollment: 150 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Adverse event reporting (Safety) | 6 months, 1 year
  Device related, procedure-related and all serious adverse events
Performance/Effectiveness - Reduction in UUI or UF episodes | 6 months, 1 year
  Demonstrate a ≥ 50% reduction in the number of UUI or UF episodes on a 3-day diary

SECONDARY OUTCOMES:
Performance/Effectiveness - Improvement in Quality of Life scoring | 6 months, 1 year
  International Consultation of Incontinence Questionnaire Overactive Bladder Quality of Life (ICIQ-OABqol): questions in each subscale are scored by a summed range of 0 to 100, with a higher score indicating better quality of life. Overall score ≥ 10 points from baseline to follow-up is indicative of a clinically meaningful improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Gita Ghadimi, OD, Study Director — Boston Scientific Corporation
Locations (13):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Urology Associates, Fairhope, Alabama
  - El Camino Health, Mountain View, California
  - Tri Valley Urology, Murrieta, California
  - University of Miami, Miami, Florida
  - Louisiana State University, New Orleans, Louisiana
  - WK Clinical Research, Shreveport, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - University Hospitals Cleveland, Cleveland, Ohio
  - Utica Park Urology, Tulsa, Oklahoma
  - Urology Partners of North Texas (UPNT), Arlington, Texas
  - Texas Oncology, Houston, Texas
  - Potomac Urology, Woodbridge, Virginia

IPD SHARING:
Plan to Share IPD: No